CLINICAL TRIAL: NCT07193381
Title: Longitudinal Assessment of Ductus Venosus Doppler Parameters and Their Association With Perinatal Outcomes in Pregnancies With Intrauterine Growth Restriction
Brief Title: Ductus Venosus Doppler in IUGR Pregnancies
Acronym: IUGR-DV
Status: Recruiting | Type: Observational
Sponsor: İlayda Gercik Arzık, MD (Other Government)
Responsible Party: Sponsor-Investigator, İlayda Gercik Arzık, MD, MD, Perinatology Specialist, Izmir City Hospital
Organization: Izmir City Hospital (Other Government)
Other Study IDs: 2025/337
Record Dates: First submitted 2025-09-13; First posted 2025-09-25 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Intrauterine Growth Restriction (IUGR)
Keywords: Ductus Venosus; Doppler Ultrasound; Neonatal Intensive Care Unit (NICU)
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- IUGR Pregnancies: Pregnant women diagnosed with intrauterine growth restriction will be followed longitudinally with serial ductus venosus Doppler assessments during the third trimester. Perinatal outcomes will be recorded until delivery and the early neonatal period.

SUMMARY:
This prospective observational cohort study aims to evaluate the relationship between ductus venosus Doppler parameters and perinatal outcomes in pregnancies complicated by intrauterine growth restriction (IUGR). Pregnant women diagnosed with IUGR will undergo longitudinal Doppler assessments of the ductus venosus during the third trimester. The Doppler indices will be correlated with perinatal outcomes, including Apgar scores, neonatal intensive care unit (NICU) admission, and perinatal mortality. The study seeks to determine whether serial ductus venosus Doppler measurements can serve as predictive markers of adverse neonatal outcomes in IUGR pregnancies.

DETAILED DESCRIPTION:
Intrauterine growth restriction (IUGR) is a major obstetric complication associated with increased risks of perinatal morbidity and mortality. Accurate assessment of fetal well-being and timely prediction of adverse outcomes are critical in the management of these pregnancies. The ductus venosus, a key component of the fetal circulation, reflects central venous pressure and cardiac function. Alterations in ductus venosus Doppler waveforms have been suggested as early markers of fetal compromise.

This prospective observational cohort study is designed to longitudinally evaluate ductus venosus Doppler parameters in pregnancies diagnosed with IUGR and to explore their association with perinatal outcomes. Pregnant women meeting the inclusion criteria will undergo serial Doppler examinations of the ductus venosus during the third trimester, performed at defined intervals until delivery.

Perinatal outcomes to be assessed include Apgar scores, neonatal intensive care unit (NICU) admission, duration of hospitalization, and perinatal mortality. By correlating longitudinal ductus venosus Doppler changes with clinical outcomes, the study aims to determine whether these parameters may serve as reliable predictors of neonatal risk in IUGR pregnancies. Ultimately, this research may provide additional evidence to support the use of ductus venosus Doppler in clinical decision-making and in the timing of delivery for growth-restricted fetuses.

ELIGIBILITY:
Inclusion Criteria:

Female participants aged 18-45 years

Singleton pregnancy

Intrauterine growth restriction (IUGR) with estimated fetal weight <10th percentile for gestational age

Gestational age ≥24 weeks at enrollment

Ability to comply with scheduled follow-up visits and Doppler examinations

Signed informed consent obtained

Exclusion Criteria:

Multiple gestations (twins or higher-order pregnancies)

Major fetal congenital anomalies

Known chromosomal abnormalities

Maternal chronic systemic diseases likely to affect fetal growth (e.g., uncontrolled diabetes mellitus, severe renal disease, severe hypertension)

Maternal infections known to impact fetal growth (e.g., TORCH infections)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women aged 18-45 years with singleton pregnancies diagnosed with intrauterine growth restriction (IUGR) will be recruited from the Department of Perinatology at Izmir City Hospital. Eligible participants will be followed with serial Doppler ultrasound examinations of the ductus venosus during the third trimester and monitored until delivery and the early neonatal period.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Composite adverse perinatal outcome (perinatal mortality, Apgar score <7 at 5 minutes, NICU admission) | From delivery until neonatal discharge (up to 28 days postpartum)
  A composite outcome including perinatal mortality, Apgar score <7 at 5 minutes, and NICU admission. The association between ductus venosus Doppler indices and this composite outcome will be analyzed.

SECONDARY OUTCOMES:
Longitudinal change (slope) of ductus venosus PI during third trimester | From study enrollment through delivery (up to 14 weeks), assessed weekly
  Rate of change per week calculated from serial weekly Doppler exams.

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Golbasi, Assistant Professor, Study Director — Izmir City Hospital
Locations (1):
- Izmir City Hospital, Izmir, Bayrakli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the dataset is limited to a single-center observational study and will only be used for publication of aggregated results.